CLINICAL TRIAL: NCT03937713
Title: A Pragmatic Randomized Comparator Trial of Eszopiclone and Brief Behavioral Therapy for Insomnia in CPAP Non Adherent Veterans With PTSD and Complex Insomnia
Brief Title: Effectiveness of Combining Behavioral and Pharmacologic Therapy for Complex Insomnia in Veterans With PTSD
Acronym: PRECEPT-D
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NURB-008-18F
Record Dates: First submitted 2019-05-01; First posted 2019-05-06 (Actual); Results first posted 2025-10-21 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Complex Insomnia
Keywords: post traumatic stress disorder; complex insomnia; cognitive behavioral therapy; eszopiclone
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Eszopiclone

STUDY DESIGN:
Intervention Model Description: A randomized comparator 1:1 to explore the comparative effectiveness of combination treatment of behavioral and pharmacological interventions with behavioral therapy alone in improving sleep quality of life, Veterans with PTSD and complex insomnia.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- BBTI plus eszopiclone (Experimental): participants randomized to the combination therapy will receive eszopiclone 2 mg orally at bedtime or placebo starting with the BBTI sessions for a period of 2 weeks in combination with 4 sessions of BBTI over 4 weeks.
  Interventions: Drug: eszopiclone; Behavioral: Brief behavioral therapy for insomnia
- Brief Behavioral Therapy for Insomnia (Active Comparator): participants randomized to BBTI will receive 4 sessions of BBTI over 4 weeks.
  Interventions: Behavioral: Brief behavioral therapy for insomnia

INTERVENTIONS:
Drug: eszopiclone — Eszopiclone is a nonbenzodiazepine benzodiazepine receptor agonists, effective for both sleep onset insomnia and sleep maintenance insomnia
  Other Names: Lunesta
  Arms: BBTI plus eszopiclone
Behavioral: Brief behavioral therapy for insomnia — BBTI is based on the core principles that are fundamental to other empirically-supported behavioral treatments of insomnia delivered over four consecutive weeks.
  Other Names: BBTI

SUMMARY:
Obstructive sleep apnea (OSA) is commonly reported in Veterans with post-traumatic stress disorder, which can potentiate symptoms of anxiety and depression, daytime symptoms and worsen nightmares. Continuous positive airway pressure (CPAP) is the most effective therapy but adherence to treatment is suboptimal. Insomnia is considered a barrier to long-term adherence. The overarching theme of the proposal is to compare the effectiveness of cognitive behavioral therapy for insomnia (CBT) plus eszopiclone, a nonbenzodiazepine hypnotic, versus CBT alone in Veterans with PTSD who are diagnosed with both OSA and insomnia, using a randomized, clinical trial, on sleep quality of life, PTSD severity, and CPAP adherence.

DETAILED DESCRIPTION:
As many as 90% of Veterans with posttraumatic stress disorder (PTSD) report nightmares and insomnia and even when nightmares are excluded, sleep disturbances are the most prevalent symptoms of PTSD with roughly 50%-70% of patients suffering from co-occurring sleep disorders. The typical sleep complaints include nightmares, distressed awakenings, nocturnal panic attacks, sleep terrors and insomnia.

While it has long been established that PTSD engenders sleep disturbances and averse clinical outcomes, current investigations indicate that disordered sleep is also a risk factor for the development of PTSD. In military personnel with combat exposure, comorbid insomnia and OSA, a condition originally labeled as "complex insomnia" has emerged as one of the most challenging sleep disorder to manage. In the presence of PTSD, the co-occurrence of OSA and insomnia is also associated with significant morbidity. Veterans with both PTSD and complex insomnia report more psychiatric symptoms, chronic pain, and higher rates of suicide. Further, these Veterans may have more difficulty adhering to CPAP because of increased awareness of the mask due to frequent awakenings and an inability to initiate or return to sleep with the mask in place. Fortunately, there are effective treatments for each of these sleep disorders. Traditional treatment models consist of treating OSA first, followed by adjunctive or concurrent treatment for insomnia only if the response to CPAP is deemed unsatisfactory. However, the suboptimal response observed in Veterans with PTSD from such an approach in terms of quality of life, PTSD symptoms, and CPAP adherence highlights the need to examine alternative modalities of treatment. At present, there are no general guidelines on the best strategy to treat complex insomnia in Veterans with PTSD. Prior studies have shown that cognitive behavioral therapy (CBT) is effective for treating insomnia when compared with hypnotic agents.Whether combination therapy offers a therapeutic advantage over CBT alone for complex insomnia in Veterans with PTSD is yet to be determined. The objective of this proposal is to conduct a pragmatic, randomized, parallel clinical trial comparing the effectiveness of Brief Behavioral Therapy for Insomnia in Military Veterans (BBTI-MV) plus eszopiclone, a non-benzodiazepine hypnotic, versus BBTI-MV alone in 52 combat-exposed Veterans with PTSD and OSA with coexisting insomnia on global sleep quality of life, PTSD symptoms, and CPAP adherence. The topic addresses several key areas of unmet needs for Veterans with PTSD and sleep disordered breathing. Among these are: 1) the association between complex insomnia and PTSD on global sleep quality of life; and 2) the effectiveness of combined treatment of CBT and eszopiclone versus CBT alone in improving sleep quality and PTSD symptoms; and 3) the impact of each treatment regimen on CPAP adherence. By establishing the most effective therapy in alleviating insomnia that complicates the presence of OSA in Veterans with PTSD, higher CPAP adherence will ultimately translate into improved cognitive function, enhanced quality of life, and suppression of PTSD symptoms. The long term benefit of this trial will also lead to opportunities for more personalized treatment including delivery method via mobile health technologies which will allow greater assimilation of results across several domains.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years and <65 years old
* Diagnosis of PTSD as determined by the intake conducted through the PTSD Clinic or the Mental Health Clinic
* Documented obstructive sleep apnea by polysomnography (AHI 5 or more/hour) who are non-adherent to CPAP as defined by device usage of less than 4 hours per night
* Chronic ( 3 months' duration) insomnia disorder
* Psychotherapeutic treatment stable for at least 4 weeks prior to randomization
* Capable of giving informed consent

Exclusion Criteria:

* Insomnia secondary to pain
* History of narcolepsy and/or cataplexy
* Treatment for seizure disorders
* Pregnant or lactating
* History of clinically significant hepatic impairment
* History of hypersensitivity, intolerance, or contraindication to eszopiclone
* Use of potent cytochrome p450 3A4 inhibitor medications (ritonavir, nelfinavir, indinavir, erythromycin, clarithromycin, troleandomycin, ketoconazole, itraconazole) and is unwilling or it is clinically contraindicated to stop the medication
* Unwilling to try or use CPAP
* Diagnosis of current schizophrenia or schizoaffective disorder
* Diagnosis of a substance dependence/abuse disorder in the past year
* History of complex nocturnal behaviors while using eszopiclone
* Severe psychiatric instability or severe situational life crises, including evidence of being actively suicidal or homicidal, or any behavior which poses an immediate danger to patient or others
* Diagnosis of bipolar disorder
* Consumption of more than two alcoholic beverages per night
* Documented or self-reported resolution of insomnia from current behavioral or pharmacological treatment of insomnia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ali A El-Solh, MD MPH, Principal Investigator — VA Western New York Healthcare System, Buffalo, NY
Locations (1):
- VA Western New York Healthcare System, Buffalo, NY, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Final de-identified data sets will be made available upon specific request and under and authorized DUA. This, in addition to the publications being made available via PubMed Central will enable validation of results by recipients.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The de-identified data will be available after the primary manuscript is published
Access Criteria: The de-identified data will be available after the primary manuscript is published for a period of 6 years

REFERENCES:
- [Derived] El-Solh AA, Lawson Y, Martinson A, Wilding G. Cognitive Behavioral Therapy Alone or in Combination with Eszopiclone in Comorbid Insomnia and Obstructive Sleep Apnea in Veterans with Posttraumatic Stress Disorder: A Randomized Trial. Psychiatr Q. 2025 Dec;96(4):787-802. doi: 10.1007/s11126-025-10143-9. Epub 2025 Apr 9. PMID 40202618

RESULTS

PARTICIPANT FLOW:
Recruitment Details: During the period extending from January 4th, 2020, and December 28th, 2023, we assessed 425 veterans with PTSD for eligibility.
Pre-assignment Details: Three hundred sixty-three Veterans were excluded because of prior treatment with CBT-I and/or active use of hypnotics (81%), presence of concurrent active medical or unstable psychiatric conditions (5%), active substance abuse (1%), documented sleep disorders other than COMISA (4%), or unable to commit for the duration of the trial (9%). Of the 62 veterans who met eligibility, nine did not meet the criteria for clinical insomnia by ISI.
Groups:
- BBTI: participants randomized to BBTI will receive 4 sessions of BBTI over 4 weeks.
  Brief behavioral therapy for insomnia: BBTI is based on the core principles that are fundamental to other empirically-supported behavioral treatments of insomnia delivered over four consecutive weeks.
Period: Overall Study
Arm/Group | BBTI Plus Eszopiclone | BBTI
Started | 26 | 27
End of Treatment | 24 (During the 6-week treatment phase, 24 completed all four sessions in the BBTI plus ESZ. Two dropped out.) | 23 (During the 6-week treatment phase, 23 completed all four sessions in the BBTI group. Four dropped out.)
End of Study | 22 (One was lost for follow-up, and one dropped out.) | 21 (Two dropped out.)
Completed | 22 | 21
Not Completed | 4 | 6
Not completed — Withdrawal by Subject | 3 | 6
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BBTI Plus Eszopiclone | BBTI | Total
Number analyzed (Participants) | 26 | 27 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.0 (7.3) | 48.4 (9.3) | 48.2 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 22 | 24 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 25 | 27 | 52
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 8 | 12
  White | 21 | 18 | 39
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 26 | 27 | 53
BMI [Mean (Standard Deviation); unit: kg.m(-2)] — Body Mass Index
  kg.m(-2) | 32.8 (6.8) | 33.0 (6.6) | 32.9 (6.7)
Pittsburgh Sleep Quality Index (PSQI) [Mean (Standard Deviation); unit: units on a scale] — Pittsburgh Sleep Quality Index. An overall score ranges from 0 to 21, where lower scores denote a healthier sleep quality.
  units on a scale | 13.0 (3.4) | 13.7 (2.7) | 13.4 (3.1)
PTSD checklist-5 (PCL-5) [Mean (Standard Deviation); unit: units on a scale] — PTSD Checklist. A total symptom severity score (range 0-80) can be obtained by summing the scores from each of the 20 items that have response options from 0 "not at all" to 4 "extremely". Higher score indicates worse symptoms.
  units on a scale | 34.5 (11.5) | 30.1 (12.8) | 32.2 (12.2)
Apnea-Hypopnea Index (AHI) [Mean (Standard Deviation); unit: events per hour] — The Apnea-Hypopnea Index (AHI) is a metric used to assess the severity of sleep apnea. It represents the number of apneas (complete cessation of airflow) and hypopneas (partial reduction of airflow) that occur per hour of sleep. The AHI is calculated by dividing the total number of apneas and hypopneas by the total hours of sleep.
  the formula for calculating AHI:
  AHI
  = Number of Apneas + Number of Hypopneas Total Sleep Time in Hours AHI= Total Sleep Time in Hours Number of Apneas + Number of Hypopneas
  events per hour | 29.2 (22.9) | 32.7 (25.3) | 31.0 (24.1)
Beck Depression Inventory (BDI) [Mean (Standard Deviation); unit: units on a scale] — The Beck Depression Inventory (BDI) is a self-report questionnaire used to assess the severity of depression. The BDI consists of 21 items, each reflecting a specific symptom or attitude related to depression.
  Each item is scored on a scale from 0 to 3, with 0 indicating the absence of the symptom and 3 indicating a severe presence of the symptom. The total score is the sum of the scores for all 21 items, and it can range from 0 to 63. Higher scores indicate a worse outcome, reflecting more severe depressive symptoms.
  units on a scale | 15.7 (8.5) | 16.1 (13.1) | 15.9 (11.1)
Insomnia Severity Index (ISI) [Mean (Standard Deviation); unit: units on a scale] — The Insomnia Severity Index (ISI) is a self-report questionnaire used to assess the severity of insomnia in adults. The ISI consists of seven items, with each item scored on a scale from 0 to 4. The total score is the sum of the scores for all seven items, and it can range from 0 to 28.Higher scores indicate a worse outcome, reflecting more severe insomnia symptoms.
  units on a scale | 18.2 (4.3) | 18.7 (4.1) | 18.3 (4.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in Pittsburgh Sleep Quality Index (PSQI) (32) at 6 Months Post-randomization
Description: The Pittsburgh Sleep Quality Index is a 19-item, self-rated questionnaire, assessed various aspects of sleep, sleep quality, and sleep disturbances. The PSQI is composed of 7 components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of scores for these 7 components yields 1 global score. An overall score ranges from 0 to 21, where lower scores denote a healthier sleep quality.
Time Frame: repeated measures between baseline and 6 months post randomization
Population: All analyses were based on the intention-to-treat principle
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | BBTI Plus Eszopiclone | BBTI
Number analyzed (Participants) | 26 | 27
units on a scale | -5.25 [-6.58 to -3.91] | -5.45 [-6.78 to -4.11]
Statistical Analysis 1: Comparison: BBTI Plus Eszopiclone vs BBTI; The sample size selected for this preliminary trial was based on the analysis of the PSQI as the primary outcome. Assuming a correlation coefficient of 0.7 between pre-and post-treatment, 21 patients per arm were needed to achieve 80% power at a significance level of 5% in order to detect a clinically significant difference of 3 units in PSQI. To compensate for an anticipated attrition rate of 25%, the recruitment target was set at 52 participants; Test type: Other — Calculations were approximated by those of a simple two-sample t-test for mean differences in PSQI in response to BBTI; p = 0.05, Mixed Models Analysis

2. Secondary Outcome: Change in PTSD Checklist-5 (PCL-5)
Description: PCL-5 is a 20-item self-report measures that have been widely used in military and civilian population to assess the severity of PTSD symptoms. A total symptom severity score (range 0-80) can be obtained by summing the scores from each of the 20 items that have response options from 0 "not at all" to 4 "extremely". Higher score indicates worse symptoms.
Time Frame: repeated measures between baseline and 6 months post randomization
Population: All analyses were based on the intention-to-treat principle
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | BBTI Plus Eszopiclone | BBTI
Number analyzed (Participants) | 26 | 27
units on a scale | -10.63 [-15.09 to -6.17] | -4.46 [-8.9 to 0.01]

3. Secondary Outcome: Change in Insomnia Severity Index (ISI)
Description: The ISI is a 7-item patient-reported outcome assessing the severity of initial, middle, and late insomnia; sleep satisfaction; interference of insomnia with daytime functioning; noticeability of sleep problems by others; and distress about sleep difficulties. The 5 point scale provides a score ranging from 0 to 28 with higher scores indicating more severe insomnia.
Time Frame: repeated measures between baseline and 6 months post randomization
Population: All analyses were based on the intention-to-treat principle
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | BBTI Plus Eszopiclone | BBTI
Number analyzed (Participants) | 26 | 27
units on a scale | -8.32 [-10.56 to -6.09] | -8.64 [-10.92 to -6.36]

4. Secondary Outcome: Change in Beck Depression Inventory-II (BDI-II)
Description: The BDI-II is a 21-item questionnaire in which respondents indicate on a four-point Likert-type scale (0=minimal to 3=severe) the presence and severity of depressive symptoms during the past 2 weeks. Items are scored on a 4-point scale ranging from 0 to 3, with higher scores indicating the presence of more depressive symptoms. The BDI-score ranges from 0 to 63. Higher scores indicate worse outcomes.
Time Frame: repeated measures between baseline and 6 months post randomization
Population: All analyses were based on the intention-to-treat principle
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | BBTI Plus Eszopiclone | BBTI
Number analyzed (Participants) | 26 | 27
units on a scale | -4.34 [-7.04 to -1.63] | -3.07 [-5.76 to -0.37]

5. Other Pre Specified Outcome: CPAP Adherence
Description: CPAP adherence will be obtained by downloading the data stored on the SmartCard. CPAP adherence is defined as the use of CPAP for 4 hours or more per night during a 28 consecutive day period. The outcome measure is the percentage of patients who met the definition of CPAP adherence based on the last 28 days prior to the 6 month time point.
Time Frame: repeated measures between baseline and 6 months post randomization
Population: All analyses were based on the intention-to-treat principle
Measure: Number; unit: percentage of participants
Arm/Group | BBTI Plus Eszopiclone | BBTI
Number analyzed (Participants) | 26 | 27
percentage of participants | 37.15 | 16.85

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | BBTI Plus Eszopiclone | BBTI
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/27
Other Adverse Events (participants affected / at risk) | 4/26 | 1/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BBTI Plus Eszopiclone (N=26) | BBTI (N=27)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Diziness (Nervous system disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-05): https://cdn.clinicaltrials.gov/large-docs/13/NCT03937713/Prot_SAP_001.pdf
  • Informed Consent Form (2020-09-23): https://cdn.clinicaltrials.gov/large-docs/13/NCT03937713/ICF_000.pdf